CLINICAL TRIAL: NCT02112279
Title: Reduction of C-Difficile Infection Using Fecal Microbiota Transplant
Brief Title: Reduction of C-Difficile Infection Using Stool Transplant
Acronym: FMT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Providence Holy Cross Medical Center (Other)
Responsible Party: Principal Investigator, Sherri Mendelson, Director Nursing Research and Magnet Program, Providence Holy Cross Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHC059
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: C-difficile
Keywords: Microbiota; c-difficile; colonoscopy; stool transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Microbiota Transplant (Experimental): Close relative or purchased donor microbiota transplant will be administered via colonoscopy; Donor microbiota applied via colonoscopy
  Interventions: Biological: Donor microbiota applied via colonoscopy.

INTERVENTIONS:
Biological: Donor microbiota applied via colonoscopy. — B. Preparation of donor sample 1. Instillation via Colonoscopy
  1. Stool mixture is administered into the terminal ileum and cecum through the biopsy channel of a colonoscope while the patient is sedated.
  Administer 300-700 ml of slurry through biopsy channel of colonoscope with a piston syringe.

SUMMARY:
Clostridium-difficile (C-difficile) is a gram positive anaerobic spore-forming bacterium that can lead to severe diarrhea and pseudomembranous colitis. According to Schroeder (2005), there are approximately 3 million cases annually with a mortality rate of 1-2.5 %. It is most often associated with overuse of antibiotics. According to Bartlett & Gerding (2008), 15-25% of anti-microbial-associated diarrhea is caused by C-difficile.

The purpose of this study is to determine if donor fecal microbiota transplant via colonoscopy reduces refractory C-difficile infection better than current routine methods such as continued antibiotic treatment. Specifically, we hypothesize that fecal microbiota transplant via colonoscopy will result in a higher C-difficile cure rate in affected patients versus care as usual in a retrospective cohort.

DETAILED DESCRIPTION:
Background

Clostridium-difficile (C-difficile) is a gram positive anaerobic spore-forming bacterium that can lead to severe diarrhea and pseudomembranous colitis. According to Schroeder (2005), there are approximately 3 million cases annually with a mortality rate of 1-2.5 %. It is most often associated with overuse of antibiotics. According to Bartlett & Gerding (2008), 15-25% of anti-microbial-associated diarrhea is caused by C-difficile.

The purpose of this study is to determine if donor fecal microbiota transplant via colonoscopy reduces refractory C-difficile infection better than current routine methods such as continued antibiotic treatment. Specifically, we hypothesize that fecal microbiota transplant via colonoscopy will result in a higher C-difficile cure rate in affected patients versus care as usual in a retrospective cohort.

Current concerns with C-difficile

An increase in C-difficile exposure in hospital settings, especially for immune compromised patients has been noted. The long life of C-difficile spores with poor ability for cleaning agents to kill the spores is a particular concern for patients in critical care and oncology units. In addition, although C-difficile has been considered a hospital acquired disease, there has been an increase in community acquired C-difficile infection with the last few years.

A concern was expressed by Muto, et al (2005) regarding the relationship between an unexpected outbreak of C-difficile infection following an increase in fluoroquinalone use. They found that exposure to levofloxacin was an independent risk factor for C-difficile-associated diarrhea and appeared to contribute substantially to the outbreak. They recommended restricted use of levofloxacin and the other implicated antibiotics to control the outbreak. In 2005 the Center for Disease Control (CDC) issued a warning regarding a new, highly toxic strain of C-difficile that was resistant to fluoroquinalone antibiotics.

A study by Sethi, et al, (2010), demonstrated the difficulty in eradicating C-difficile infections. In their study of fifty-two patients with C-difficile, the bacteria were suppressed to undetectable levels in stool samples from most patients during treatment. At 1-4 weeks after treatment, 56% of patients who had samples tested were asymptomatic carriers of C-difficile. They found that skin contamination and environmental shedding of C-difficile often persist at the time of resolution of diarrhea, and recurrent shedding is common 1-4 weeks after therapy (58% for skin contamination and 50%, for environmental shedding).

Treatment with fecal microbiota Microbiotas are friendly, beneficial bacteria. Microbiotas produce essential nutrients such as short-chain fatty acids; control epithelial cell growth; prevent overgrowth of infectious organisms; boost intestinal immunity; and prevent inflammation, diarrhea and other intestinal conditions. This essential ecosystem provides an important balance between health and disease in the body. The goal for fecal microbial transplant is to re-establish fecal microbial homeostasis with increased microbial diversity.

Fecal microbiota transplants are a relatively new direction in treating C-difficile infections (CDI) that are refractory to accepted antibiotic treatment. In a retrospective medical record review of 70 patients with recurrent CDI who had undergone fecal transplantation performed via colonoscopy, Matilla, et al (2011) concluded that fecal transplantation through colonoscopy seems to be an effective treatment for recurrent CDI and also for recurrent CDI caused by the virulent C-difficile 027 strain.

According to a systematic review of the literature, in 317 patients treated across 27 case series and reports, intestinal microbiota transplant demonstrated disease resolution in 92% of cases. Among the variables that determined procedural success were treatment prior to procedure, relationship of the donor to the patient, route of fecal microbiota instillation and amount of fecal microbiota solution delivered. (Gough, Shaikh & Manges, 2010).

A three-group study was conducted with 13 participants randomized to each group. Results demonstrated resolution rates of C-difficile were (81%) for the vancomycin group with subsequent donor fecal transplant via nasoduodenal tube; (31%) vancomycin only group; and (23%) vancomycin with bowel lavage group; p<0.0001 (van Nood, et al; 2013).

In a published report of proceedings of a Canadian Working Group to discuss the issues of fecal microbiota transplant, many important concerns were brought forward, including the need for donor screening, standardization of the donor fecal transplant material and the use of biologic material as an un-approved drug (Allen-Vercoe, et al, 2012). These issues must be addressed in any study to ensure that patient safety and study reliability are at the forefront in the determination of the effectiveness of fecal transplant to treat C-difficile infections that are refractory to approved antibiotic treatment.

Methods

This study is a one-group convenience sample interventional study with a qualitative component.

Recruitment Active recruitment will involve one-to-one explanations with in-patients at a community hospital and out-patients presenting one of the study physicians for care of refractory C-difficile infection.

Procedures I. Participants

A. Patient:

1. Patients must be 18 years of age or older
2. Patient must have a positive C. difficile test within the 10 days prior to the procedure.
3. Continued symptoms of c-difficile infection
4. Patients must have failed at least two courses of appropriate antibiotic therapy for C. diff to be a candidate for this procedure.
5. Informed consent must be obtained.
6. All antibiotics must be discounted at least 72 hours prior to the infusion. The patient may continue on proton pump inhibitors (PPIs) but their use should be noted pre- and post- transplant.
7. A standard colonoscopy prep will be given the day before the procedure (Laxative regimen and clear liquids only).
8. Patient must provide a clean, dry blender that will be used to blend the stool mixture. The blender will be discarded after use and will not be re-used.

B. Donor: if Familial versus purchased donor stool

1. The donor must be 18 years of age or older.
2. The closer the relationship between the donor and the recipient the better. Spouses and partners, first degree relatives, or household members are preferred.
3. Donors must have no history of Hepatitis B or C, HIV, recent communicable disease, incarceration, high-risk sexual behavior, inflammatory bowel disease, gastrointestinal malignancy or colon polyps. They may not have traveled an area known to be endemic for diarrheal illnesses in the past 6 months, taken antibiotics in the past 3 months for any reason, or be on any immunosuppressive drugs or chemotherapy.
4. Donors must test negative for Hepatitis B and C and HIV, and have stool specimens negative for C. Difficile, Campylobacter, Salmonella, Shigella, ova and parasites, other pathogenic bacteria, giardia antigen and cryptosporidium antigen within 10 days prior to the procedure.
5. Informed consent must be obtained from the donor.

II. Setting A. A Gastroenterology Laboratory in an acute care 377-bed non-teaching hospital.

III. Procedure A. Prior to Procedure

1. Verify physician order for Bowel Recolonization Therapy (or Fecal Bacteriotherapy) via colonoscopy.
2. Stool from donor must be brought in to the hospital in an approved container, received by hospital staff, labeled with the donors name, the recipients name and the recipients medical record number and sent to Endoscopy for preparation for procedure.

   a) The stool from donor should be formed and of adequate quantity. b) The stool from donor should be collected as close in time to instillation as possible, preferably within 6-8 hours of the procedure.
3. Informed consent must be obtained from the donor and the recipient. B. Preparation of donor sample

<!-- -->

1. Personal protective equipment (mask, eye protection, gown and gloves) must be worn throughout the preparation procedure
2. Blend stool and non-bacteriostatic normal saline in a blender until stool reaches a liquid slurry consistency. Add more non-bacteriostatic normal saline until desired consistency achieved. The stool should be blended to the approximate consistency of a milkshake.
3. Filter stool solution into a sterile container with 6 layers of gauze pads, removing as much particulate matter as possible
4. Large volumes of 300-700 ml should be used for delivery through the colonoscope into the cecum or terminal ileum.
5. Container with fecal slurry must be labeled with recipients identification information and delivered immediately to bedside for instillation.

C. Instillation via Colonoscopy

1. Stool mixture is administered into the terminal ileum and cecum through the biopsy channel of a colonoscope while the patient is sedated.

1. Equipment:

   (1) 5 syringes (at least 60 cc each) (2) K-Y jelly or water-soluble lubricant (3) Chux pads (4) Exam gloves
2. Complete hand hygiene.
3. Verify correct patient by using two patient identifiers.
4. Put on gloves and place a drape/chux under the patients buttocks.
5. Administer 300-700 ml of slurry through biopsy channel of colonoscope with a piston syringe.
6. Dispose of any leftover slurry into toilet. Dispose of waste.
7. Remove gloves and complete hand hygiene.
8. Document

   1. Date and time of procedure
   2. Amount of fecal slurry administered.
   3. Results and patients response to procedure.
   4. Observe patient for at least 15-30 minutes, until VS are stable.

   Measurement and data collection
   1. All study patients will keep a stool diary for the 30 days following the transplant noting number of stools, time of passage, character of stool, and any changes in the patients quality of life.
   2. All study patients will have a C. difficile toxin determination test at 14 days and 28 days after the procedure per physician order. C. difficile testing may be conducted using one of three methods: PCR, Illumegene, or EIA.
   3. Recurrence of C. difficile is determined by C. difficile tests, signs and symptoms, as well as the consistency of stools produced.
   4. Study patients will be contacted at 7, 14 and 28 days following the procedure for any concerns. A self-addressed envelope will be provided to the study participants to return their completed post-procedures log to the research team after 28 days.
   5. Records for patients who undergo this procedure will be maintained by the research team in a secure location.

      Analysis Data analysis will be completed using measures of central tendency and raw percentages. Results of the post-procedure phone calls and the patient logs will be analyzed using qualitative measures based on phenomenology and measures of central tendency for quantitative aspects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older
2. Patient must have a positive C. difficile test within the 10 days prior to the procedure
3. Continued symptoms of c-difficile infection
4. Patients must have failed at least two courses of appropriate antibiotic therapy for C. diff to be a candidate for this procedure

   -

Exclusion Criteria:

1. Under 18 years of age
2. Negative C. difficile test within the 10 days prior to the procedure
3. No symptoms of c-difficile infection
4. Less than two courses of appropriate antibiotic therapy for C. difficile infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Negative c-difficile test | 30 days
  Enrolled patients will test negative for c-difficile following application of the study intervention

SECONDARY OUTCOMES:
Relief of symptoms | 30 days
  patient report of decrease in symptoms related to c-difficile

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Moghimi, MD, Principal Investigator — PHCMC; Ellsworth Pryor, MD, Principal Investigator — Providence Holy Cross Medical Center; Sherri G Mendelson, RN, PhD, Principal Investigator — Providence Holy Cross Medical Center
Locations (1):
- Providence Holy Cross Medical Center, Mission Hills, California, United States